CLINICAL TRIAL: NCT04421261
Title: Evaluation of Performance of Air-Q Self Pressurized Airway Device With Blocker and Proseal Laryngeal Mask Airway at Different Head and Neck Positions in Anesthetized Paralyzed Adult Female Patients Undergoing Elective Gynecological Operations
Brief Title: Ventilation With Supraglottic Airway Devices
Status: Completed | Type: Observational
Sponsor: Reham Ali Abdelhaleem Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Reham Ali Abdelhaleem Abdelrahman, Anesthesia lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: KR-1990
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Laryngeal Masks Comparison

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Air-Q Self Pressurized Airway Device with Blocker
  Interventions: Device: Air-Q Self Pressurized Airway Device with Blocker
- Proseal Laryngeal Mask Airway
  Interventions: Device: Proseal Laryngeal Mask Airway

INTERVENTIONS:
Device: Air-Q Self Pressurized Airway Device with Blocker — used in low risk adult females undergoing elective surgeries
  Groups: Air-Q Self Pressurized Airway Device with Blocker
Device: Proseal Laryngeal Mask Airway — used in low risk adult female patients undergoing elective surgeries
  Groups: Proseal Laryngeal Mask Airway

SUMMARY:
Airo-Q Self Pressurized airway device with Blocker will be compared with Proseal LMA in anesthetized adult female patients undergoing elective surgeries to discuss the influence of different head and neck positions on the performance of both devices. Oropharyngeal leak pressure, peak inspiratory pressure, ventilation score and fiber-optic view will be assessed in neutral, flexion, extension and lateral positions in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients ASA I&II.
* age: 18-55 years old.
* BMI< 35.
* undergoing elective surgeries.

Exclusion Criteria:

* Patients with history of upper respiratory tract infections and obstructive sleep apnea.
* Patients who are potentially full stomach such as trauma, pregnancy, history of gastric regurgitation &heart burn, those with esophageal reflux or hiatus hernia.
* Patients with coagulation disorders.
* Patients with El-Ganzouri airway score ≥ 5 will.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult female patients who will be admitted through outpatient clinic of Kasr alainy hospitals
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
oropharyngeal leak pressure | 1 year
  pressure at which air leak starts to occur

CONTACTS AND LOCATIONS:
Locations (1):
- Department of anesthesia, Surgical ICU and Pain Management, Cairo, Egypt